CLINICAL TRIAL: NCT06900621
Title: Effects of Two Different Methods on Early Period Dry Mouth After Septoplasty Surgery
Brief Title: Effects of Methods on Dry Mouth After Septoplasty Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, dürdane palabıyık yılmaz, PhD Student, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EGE-SBE-DPY-01
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Septoplasty; Dry Mouth
Keywords: dry mouth; nursing; early period; septoplasty; water at room temperature; ice water
MeSH Terms: conditions — Xerostomia | interventions — major intrinsic protein, plant

STUDY DESIGN:
Intervention Model Description: This study was planned as an experimental, randomized controlled, single-blind study.Patients who meet the postoperative criteria will be randomized to one of three groups. Randomization was performed as a 3-way block randomization (Sealed Envelope Ltd. 2022). In the study, 3-way block randomization was applied using a blind technique. 3 participants in each block were assigned to different groups in a randomized order. The group codes determined in accordance with the randomization list were used to assign participants to the experimental conditions. This randomization method was preferred in order to provide balance between the participant groups and to minimize the potential effects of external factors.
Who Masked: Participant
Masking Description: The instructions given to the participants during the application process were designed in line with the blinding principles and aimed to prevent information leakage regarding which group the participants belonged to. During the data collection phase, the group information of the participants was recorded, but this information was not used during the analysis phase, ensuring that the blinding status was maintained. For blinding, a separate envelope containing each block code was prepared and a unique code indicating which block it belonged to was added to each envelope. The blocks were arranged in a randomized order and the envelopes belonging to each block were arranged according to this order. This process ensured that the participants in each block were randomly assigned to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ice Water (Group 1) (Active Comparator): Patients who come to the surgical clinic after the surgery will be given a VAS score for dry mouth at the 30th minute. Immediately afterwards, 5 ml of ice water (5-9 °C) placed in spray cans every 30 minutes will be sprayed into the mouth, tongue, palate, floor of the mouth, inside the right and left cheeks until all the water is used up. This application will be applied to the intervention groups a total of 5 times (30th min-60th min-90th min-120th min-150th min). VAS scoring will be done for dry mouth before each application. The first oral intake of the patients is routinely started at the 180th minute. After the applications are completed, VAS scoring will be requested for the satisfaction evaluation of the patients in the intervention group.
  Interventions: Other: ice water
- Room Temperature Water (Group 2) (Active Comparator): Patients who come to the surgical clinic after the surgery will be given a VAS score for dry mouth assessment at the 30th minute. Immediately afterwards, 5 ml of room temperature water (15-24 °C) placed in spray cans every 30 minutes will be sprayed into the mouth, tongue, palate, floor of the mouth, inside the right and left cheeks until all the water is used up. This application will be applied to the intervention groups a total of 5 times (30th min-60th min-90th min-120th min-150th min). VAS scoring will be done for dry mouth before each application. The first oral intake of the patients is routinely started at the 180th minute. After the applications are completed, VAS scoring will be requested for the satisfaction assessment of the patients in the intervention group.
  Interventions: Other: room temperature water
- Control (Group 3) (No Intervention): The routine application in the clinic (oral intake restriction for 3 hours after surgery) will be applied to the control group. No application will be made, dry mouth will be evaluated at the specified times.

INTERVENTIONS:
Other: ice water — Patients who apply SPTM are given a semifowler position with the head of the bed at least 45°, if there is no contraindication. The water temperature (5-9 °C) will be measured with a calibrated digital thermometer. After VAS scoring, patients are sprayed with 5 ml of ice water placed in spray cans every 30 minutes until all the water is used up in the mouth, tongue, palate, floor of the mouth, inside the right and left cheeks, depending on the group. A total of 5 rounds are made with 5 ml of water in one round (0.2 ml is sprayed on the tongue, palate, floor of the mouth, inside the right and left cheeks) and each round is planned to be completed in 1 minute and last at most 5 minutes. This application is applied to the intervention groups 5 times in total (30th min- 60th min- 90th min- 120th min- 150th min). The first oral intake of the patients is routinely started at the 180th minute.
  Arms: Ice Water (Group 1)
Other: room temperature water — Patients who apply SPTM are given a semifowler position with the head of the bed at least 45°, if there is no contraindication. The water temperature (15-24 °C) will be measured with a calibrated digital thermometer. After VAS scoring, patients are sprayed with 5 ml of room temperature water placed in spray cans every 30 minutes until all the water is used up in the mouth, tongue, palate, floor of the mouth, inside the right and left cheeks, depending on the group. A total of 5 rounds are made with 5 ml of water in one round (0.2 ml is sprayed on the tongue, palate, floor of the mouth, inside the right and left cheeks) and each round is planned to be completed in 1 minute and last at most 5 minutes. This application is applied to the intervention groups 5 times in total (30th min- 60th min- 90th min- 120th min- 150th min). The first oral intake of the patients is routinely started at the 180th minute.
  Arms: Room Temperature Water (Group 2)

SUMMARY:
It was planned to investigate the effects of two different methods on early dry mouth after septoplasty surgery. The data of this study, which is planned to be conducted experimentally, is planned to be collected at Gönen State Hospital between 2025-2026. Patients who are scheduled to undergo septoplasty surgery and present with septum deviation constitute the universe of the study. The research sample (n: 63) was determined using the Power analysis G*Power v3.1.9.7 program by taking the sample study as reference. However, considering the data losses (dropouts) in similar studies, when the missing data rate was taken as 20% , the sample size was determined as 81 patients. Patients who were informed about the study and volunteered to participate in the study (n: 81) and met the inclusion criteria of the study will constitute the sample group. 3 groups were determined in the study as intervention groups (group 1 and group 2) and control group (group 3). Patients who meet the preoperative criteria will be randomized into one of three groups after surgery. Data will be collected using the Patient Identification Form, General Patient Follow-up Form, Nasal Obstruction Symptom Assessment Scale (NOSE), Visual Analog Scale (VAS) scoring expressed by the patient to measure mouth dryness and satisfaction, "Safety Protocol for Thirst Management in the Immediate Postoperative Period" (SPTM), Oral Mucous Membrane Integrity Assessment and Follow-up Form - Oral Assessment Guide (OAG). 3 groups will be created in the study. 5 ml of ice water will be applied to one group that will receive intervention, the other group will be given water at normal room temperature, and the control group will receive standard clinical care and will not be treated. As a result of the evaluation made with SPTM in the first 30 minutes after the surgery, the dry mouth of all patients included in the study (Group 1, Group 2, Group 3) who meet the conditions will be evaluated before the application, starting from the first 30 minutes after the surgery and at 60 - 90 - 120 - 150 - 180 minutes. In the study, all patients (Group 1, Group 2, Group 3) will be evaluated for dry mouth before the application. The data obtained as a result of the study will be analyzed with a statistical package program. In the evaluation of the data in the study, descriptive statistics and parametric or non-parametric tests will be applied depending on whether the data show a normal distribution. In comparisons, p<0.05 value will be considered statistically significant.

DETAILED DESCRIPTION:
Nasal septum deviation (NSD) is one of the most common upper respiratory tract diseases causing airway obstruction, with some authors reporting a prevalence of up to 70-80% in the general population. In NSD, breathing through the mouth instead of the nose may cause complaints of dry mouth and sore throat. In addition to NSD, diseases and medications that cause dry mouth include the presence of an endotracheal tube in intensive care patients, the presence of an orogastric or nasogastric tube, frequent oral aspiration, therapeutic dehydration (e.g. cardiogenic shock or ARDS), not taking fluids or nutrients by mouth, fever, diarrhea, burns, continuous oxygen therapy, dysphagia, fear, and anxiety. Klavuz et al. (2022) found that gender did not have much of an effect on dry mouth and the prevalence of dry mouth could be seen at different rates as a result of their study conducted between the ages of 16-90. In addition, it was observed that smoking reduced the salivary flow rate; however, it was not the primary factor causing hyposalivation. Although septoplasty is the most commonly performed surgery in NSD, the severity, side and type of nasal obstruction should be taken into consideration when making the surgical decision. Özkiriş and Mutlu (2010) stated that NSD was determined in 39% of 20,596 patients and only 2,113 of the patients had complaints of nasal obstruction and surgery was applied to approximately 55% of them. The terms dry mouth and thirst, which are often used interchangeably, are the most common symptoms of terminal dehydration, along with nausea, vomiting and fatigue. The patient's feeling of dry mouth is defined as a distressing discomfort. Preoperative fasting, medication use during anesthesia-surgery, mechanical ventilation with an endotracheal tube, application of devices such as airway, blood loss during surgery, etc. may present situations that encourage and increase the appearance of thirst, and may also cause deterioration of oral health, salivary flow rate and content in patients. Moon et al. (2015) compared cold water and cold saline gauze in their study and concluded that wet gauze can be applied with cold normal saline to reduce thirst and salivary acidity and improve the condition of the oral cavity in patients after surgery. Thirst and dry mouth increase as decreased salivary flow decreases the pH of saliva. The risk of dry mouth is defined as sensitivity to discomfort or damage in the oral mucosa due to decreased quantity or quality of saliva, while mouth breathing is among the risk factors for the diagnosis of oral mucous membrane deterioration. In the literature, it is stated that sipping a small amount of water is the most common and practical method in the treatment of dry mouth; in addition, mouthwashes, moisturizing products and artificial saliva products are effective in improving the quality of life and maintaining and protecting oral health. Many different methods have been used for the intervention of postoperative dry mouth before and after surgery. Garcia (2019) reported that in the preoperative application of mentholated chewing gum, dry mouth increased from 64.7 to 72.5 in the control group and decreased from 64.7 to 3.9 in the intervention group. In a similar study, dry mouth also decreased. In bariatric surgery patients in the PACU with videolaparoscopy, the use of a mentholated pack was not more effective than a non-mentholated precaution pack in terms of reducing thirst intensity, improving lip hydration, dryness and oral cavity taste for one hour, and the mentholated strategy was proven to be effective after a single application. In a similar study, it was found that a mentholated care pack only improved the tongue and saliva in postoperative patients undergoing abdominal surgery. In the study of Oztas and Oztas (2022), no significant difference was found between the three groups in terms of age, gender, ASA, preoperative thirst and dry mouth, and preoperative oral health status. A significant difference was found between the groups after 8, 20, 24, 36, and 40 hours in terms of thirst and dry mouth severity scores. The intervention group receiving cold water spray showed statistically significant differences when compared with the control groups receiving cold saline and 1-2 ml room temperature water, but no significant difference was found between the oral health status and pH scores after 4, 8, 20, 24, 36, and 40 hours. It shows that cold water spray is more effective on the thirst and dry mouth scores of patients undergoing major abdominal surgery compared to cold normal saline spray and water applied using a syringe, but it is not an effective factor on oral health status and saliva pH values. Hur et al. (2009) examined the effects of gargling with cold water, applying wet gauze and moisturizing after nasal surgery; a significant decrease in mouth dryness was found in the intervention group at 2-4 hours, and a significant decrease in mouth dryness was found in the control group at 4 hours. As a result, gargling with cold water was found to be an effective nursing intervention to reduce postoperative thirst and dry mouth, and gargling with cold water was found to be effective in reducing thirst in relation to the duration. Gu et al. (2022) compared wiping with cold water gauze and not wiping with cold water gauze in patients undergoing nasal surgery, and concluded that there was no significant difference between the two groups in terms of thirst and oral status after the intervention, but thirst and oral status improved significantly. However, no study has been found that evaluates the effects of ice water and room temperature water interventions on dry mouth after septoplasty surgery. The subject of this thesis is to examine the effects of interventions on dry mouth in patients after septoplasty. The aim of this study is to investigate the effects of two different methods on early period dry mouth after septoplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 89
* Able to communicate in Turkish
* No obstacle to communication
* Agreeing to participate in the study
* Conscious and oriented as a result of the evaluation made with SPMT at 30 minutes after the surgery, with a clear airway, no nausea or vomiting
* Using silicone nasal tampons

Exclusion Criteria:

* Patients with a preoperative oral mucous membrane integrity assessment Oral Assessment Guide (OAG) result of over 16
* Those taking medication that affects dry mouth
* Those with a chronic disease that affects dry mouth
* Those undergoing a second simultaneous surgical procedure
* Those who develop complications during surgery and/or during recovery from anesthesia
* Patients who smoke will not be included in the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
dry mouth | The evaluation of dry mouth with VAS will be done once before the surgery and 6 times after the surgery and will take a total of 3-5 minutes.
  Pre-Operative: Patients will be checked in terms of inclusion and exclusion criteria in the clinic and if they are suitable, they will be asked to participate in the study. The oral assessment guide (OAG) will be applied at this stage of the study. Patients who score 16 points or less in the OAG assessment (by the researcher using a light source and abeslang) will be included in the study. Before surgery, patients will be asked to fill out the Patient Identification Form. Then, the Nasal Obstruction Symptom Assessment Scale and the VAS scoring, expressed by the patient to measure dry mouth, will be performed and recorded in the general patient follow-up form. Post-operatively: starting from the first 30 minutes after the operation, and at 60-90-120-150-180 minutes, all patients included in the study (Group 1, Group 2, Group 3) will be evaluated for dry mouth before the application. Visual Analog Scale (VAS) will be used to determine dry mouth.

SECONDARY OUTCOMES:
patient satisfaction | Patient satisfaction evaluation with VAS will be done after the application is completed only for Group 1 and Group 2 after the operation. It will take a maximum of 1 minute.
  In the literature, VAS has been used to evaluate postoperative dry mouth (Oztas and Oztas 2022; Serato et al. 2019). VAS has also been used in the assessment of satisfaction (Oztas and Oztas 2022; Lee et al. 2020; Elmashad and Gouda, 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Eda Dolgun, Ass. Prof., Study Director — Ege University
Locations (1):
- Gönen State Hospital, Balıkesir, Gönen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No